CLINICAL TRIAL: NCT01145235
Title: Swedish Macrolane Registry
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 31GB0905
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2018-08

CONDITIONS: Breast Augmentation
Keywords: Breast augmentation with Macrolane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Females previously treated with Macrolane in their breasts.

SUMMARY:
A Registry to monitor long term safety in female subjects after treatment with Macrolane VRF20 and/or MacrolaneT VRF30 in the breasts.

ELIGIBILITY:
Inclusion Criteria:

1. Females previously treated with Macrolane VRF in the breasts
2. Females continuously being treated with Macrolane VRF in the breasts, initial treatment or re-treatment.

Exclusion Criteria:

No exclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All clinics treating females with Macrolane in the breast will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
To document the incidence of breast cancer in female subjects after treatment with Macrolane VRFs in the breasts when the product is used in clinical practice. | 2010-2015

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Per Hedén, Stockholm, Sweden